CLINICAL TRIAL: NCT05401500
Title: ACTA2 and Familial Aortopathies: Creation and Validation of an Exploratory Cellular Model
Brief Title: Familial Aortopathies and Cellular Exploration
Acronym: FACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RCAPHM22_0100
Record Dates: First submitted 2022-05-19; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Familial Aortopathies
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- familial aortopathy (Experimental)
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — blood sampling

SUMMARY:
The prevalence of hereditary aortic disease (HTAD), responsible for aneurysm or dissection, is estimated at 25%. Mutations in the ACTA2 gene represent the main cause of non-syndromic forms (10-21%). ACTA2 is expressed in vascular wall smooth muscle cells (VSMC) and encodes alpha actin (α-SMA). This actin isoform is in the majority in VSMCs and plays a key role in their contractile properties. The mutations are dominant-negative and lead, in a fibroblast model, to defects in the organisation of the actin cytoskeleton and to an increase in the migratory and proliferative potential of the cells. In vivo, VSCMs exist in a phenotypic continuum ranging from a quiescent differentiated contractile state to a so-called synthetic state in which cells are proliferative, synthesise extracellular matrix elements and exhibit enhanced migratory capabilities. To understand how ACTA2 mutations deregulate VSMC functions and steer them towards a synthetic phenotype, it is necessary to have a cellular model as close as possible to the affected tissue..

ELIGIBILITY:
Inclusion Criteria:

* patient with a mutation in the ACTA2 gene

Exclusion Criteria:

* patient under 18 years of age at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
analysis of the impact of ACTA2 mutations on the morphology of the actin cytoskeleton | baseline
  use of a model of IPS cells reprogrammed into VSMCs from patients with ACTA2 mutations, compared to a healthy control

CONTACTS AND LOCATIONS:
Overall Officials: François Cremieux, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No